CLINICAL TRIAL: NCT07381348
Title: Determination of Metabolomic Profile Differences in Possible Sarcopenia Accompanying Fibromyalgia Syndrome in Women
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Emre Adıgüzel, Emre Adıgüzel, Associate professor, Ankara City Hospital Bilkent, Ankara City Hospital Bilkent
Other Study IDs: 10025132
Record Dates: First submitted 2025-11-23; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia; Sarcopenia
Keywords: Fibromyalgia; Sarcopenia; Metabolom
MeSH Terms: conditions — Fibromyalgia; Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — blood serum metabolom analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fibromiyalgia and probable sarcopenia
- Fibromyalgia and no probable sarcopenia
- Healthy

SUMMARY:
The goal of this observational study is to determine the serum metabolome profile differences in the presence of possible sarcopenia in patients with fibromyalgia and to compare them with healthy individuals. In this way, it is aimed to contribute to the knowledge about the pathophysiology, diagnosis and treatment of these diseases.The main questions it aims to answer are:

* Is there a difference in blood metabolite levels and metabolic pathways in fibromyalgia syndrome and possible sarcopenia accompanying fibromyalgia syndrome?
* Based on these identified differences, can biomarkers be determined for these diseases?

DETAILED DESCRIPTION:
After being informed about study and potential risks, all patient giving written informed consent will undergo screening period determine eligibility for study entry. Participants will be divided into three groups: those with fibromyalgia syndrome and probable sarcopenia, those with fibromyalgia syndrome and no probable sarcopenia, and healthy people. Presence of probable sarcopenia and sarcopenia will be determined by using SARC-F scale, hand grip strength measurement with hand dynamometer, muscle mass measurement with Bioimpedance Analysis, anthropometric measurement, walking speed measurement in patients with fibromyalgia diagnosis.The serum metabolome profiles of the three groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Being between 18-60 years old
2. Being diagnosed with Fibromyalgia according to ACR 2016 diagnostic criteria
3. Having agreed to participate in the study
4. Healthy controls
5. Being a woman

Exclusion Criteria:

1. Those who cannot take command due to cognitive dysfunction
2. Pregnancy
3. Those with severe cardiac disease, COPD, malignancy, neuromuscular disease, inflammatory rheumatic disease and organ failure
4. Those with orthopedic disorders that may cause limitation in joint range of motion and/or loss of motor muscle strength
5. Patients using systemic glucocorticoid, ACE-I / ARB, statin, sulfonylurea, allopurinol

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Forty-four female patients aged 18-60 years and 22 healthy female controls who applied to the physical therapy outpatient clinics of Ankara City Hospital FTR hospital and were diagnosed with Fibromyalgia according to the American Rheumatology Society (ACR) 2016 diagnostic criteria.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Comparison of serum metabolite concentrations between groups. Plasma samples were collected from all participants. Samples were centrifuged at 1500 rpm for 10 minutes and stored at -80 degrees to be used in metabolome analysis. | through study completion, an average of 1 year
  Assesment of serum metabolite concentrations using gas chromatography/mass spectroscopy (GC/MS).
  The obtained GC/MS data were evaluated on the MS-DIAL metabolomics platform. Untargeted metabolomics studies have been conducted. Metabolites with a match score of 70 and above were accepted using the Kovats retention index database. In the pre-data analysis processes within the MS DIAL platform, peak identification, deconvolution and data alignment processes were primarily carried out. After comparing the metabolome data between the three groups, cluster analysis was performed and pathway differences between the groups were revealed. The results were evaluated at the 95% confidence interval and the significance level was p<0.05.

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | Baseline (Day 0)
  A self-administered instrument used to measure the health status of patients with fibromyalgia. Scores range from 0 to 100, where higher scores indicate a greater impact of the syndrome on the patient's life.
  Units on a scale
Hand Grip Strength measured by Hand Dynamometer | baseline
  Assessment of upper extremity muscle strength using a hydraulic hand dynamometer (e.g., Jamar). Participants perform three trials with the dominant hand, and the maximum value is recorded.
  Unit of Measure: Kilograms (kg)
Skeletal Muscle Mass Index (SMI) measured by Bioimpedance Analysis (BIA) | Baseline
  Estimation of skeletal muscle mass using a multi-frequency BIA device. The Skeletal Muscle Index (SMI) is calculated by dividing the appendicular skeletal muscle mass by the square of the height (kg/m²).
  Unit of Measure: kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Emre Adıgüzel, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital Physical Treatment and Rehabilitation Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participants did not want their personal information to be shared.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT07381348/Prot_SAP_000.pdf